CLINICAL TRIAL: NCT01504503
Title: Open Label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Oral Bioequivalence Study of Donepezil Hydrochloride Tablets 10mg With ARICEPT® (Containing Donepezil Hydrochloride) Tablets 10 mg in Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study for Donepezil Hydrochloride 10 mg Tablets Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 645/09
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Donepezil; crossover
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil Hydrochloride10 mg Tablets (Experimental): Donepezil Hydrochloride 10 mg Tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Donepezil Hydrochloride
- Aricept 10 mg Tablets (Active Comparator): Aricept 10 mgTablets of Pfizer Inc
  Interventions: Drug: Aricept

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Donepezil Hydrochloride Tablets 10 mg
  Other Names: Aricept 10 mg
  Arms: Donepezil Hydrochloride10 mg Tablets
Drug: Aricept — Aricept 10 mg Tablets
  Arms: Aricept 10 mg Tablets

SUMMARY:
This is an open label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
The study was an open label, balanced, randomized, two-treatment, two-period, two sequence,single dose, crossover, oral bioequivalence study of Donepezil Hydrochloride tablets 10 mg of Dr. Reddy's Laboratories Limited, India comparing with that of ARICEPT® (containing Donepezil Hydrochloride) tablets 10 mg of Pfizer Inc, New York, 10017 in healthy, adult, human subjects under fasting condition. 28 subjects are enrolled in the study, and 26 subjects are completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Must be healthy, adult, human beings within 18 and 45 years of age (both inclusive) weighing at least 50 kg.
* Having a body mass index between 18.0 and 24.9 (both inclusive), calculated as weight in Kg/height in m2.
* Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician / investigator to be of no clinical significance).
* Female Subjects

  * Of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

* Incapable of understanding the informed consent.
* Systolic blood pressure less than 90 mm of Hg 140 mm of Hg.
* Diastolic blood pressure less than 60 mm of Hg 90 mm of Hg.
* Oral temperature is below 95.0°F or above 98.6°F.
* Pulse rate below 50/min or above 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Consumption of grapefruit for the past ten days prior to the check-in, in each period.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.
* Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period.
* Difficulty in abstaining from xanthene containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period.
* Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing.
* Clinically significant abnormalities and / or with significant diseases.
* Confirmed positive in alcohol screening.
* Confirmed positive in selected drug of abuse.
* Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
* Confirmed positive in urine pregnancy test.
* Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Area unde curve (AUC) | Pre-dose 0.5,0.75,1,1.5,2,2.5,3,3.5,4,4.5,5,5.5,6,7,8,9,10,12,16,24,36,48,72,96,120,144,168,192,216,240 and 264 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. L Krishna Murthy, Principal Investigator — Bioserve Clinical Research Private Limited
Locations (1):
- Bioserve Clinical Research Private Limited, Hyderabad, Andhra Pradesh, India